CLINICAL TRIAL: NCT07388758
Title: Efficacy and Safety of Scipibaimab Combined With Tislelizumab in the Treatment of Patients With Recurrent and Metastatic Nasopharyngeal Carcinoma Who Have Failed First-line Treatment: a Multicenter, Single-arm, Non-randomized, Open-label Phase II Clinical Study
Brief Title: Scipibaimab Combined With Tislelizumab in Patients With First-Line Treatment-Failed Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Sichuan Cancer Hospital and Research Institute (Other); Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-070
Record Dates: First submitted 2026-01-26; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scipibaimab combined with Tislelizumab (Experimental): Patients with recurrent or metastatic nasopharyngeal carcinoma who have progressed after first-line platinum-based chemotherapy plus PD-1 inhibition will receive scipibaimab 300 mg subcutaneous and tislelizumab 200 mg intravenous every 3 weeks until disease progression, unacceptable toxicity, or completion of 2-year treatment window.
  Interventions: Drug: Tislelizumab; Drug: Scipibaimab

INTERVENTIONS:
Drug: Tislelizumab — Anti-PD-1 targeted immunotherapy
Drug: Scipibaimab — Scipibaimab (CM310) is a humanized IgG4 monoclonal antibody that selectively binds to a unique epitope on human IL-4Rα, thereby simultaneously blocking IL-4 and IL-13 signaling without competing with dupilumab's binding site; it exhibits cross-species reactivity (human, cynomolgus monkey, rat), displays linear pharmacokinetics with an estimated terminal half-life of ~300 h in monkeys, and has shown favorable safety and dose-proportional exposure in multiple Phase 1-3 trials for type-2 inflammatory diseases .

SUMMARY:
This study aims to explore the efficacy and safety of scipibaimab combined with tislelizumab in patients with recurrent or metastatic nasopharyngeal carcinoma who have progressed after first-line therapy.

DETAILED DESCRIPTION:
In the immunotherapy era, patients with recurrent/metastatic nasopharyngeal carcinoma who progress after both platinum-based chemotherapy and PD-1 blockade lack further standard options. IL-4Rα inhibition can overcome PD-1 resistance by re-activating CD8+ T cells; combining scipibaimab (anti-IL-4Rα) with tislelizumab (anti-PD-1) has shown additive activity without overlapping toxicity. This trial will assess the efficacy and safety of the combination in patients who have failed prior platinum and PD-1 therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed with recurrent or metastatic nasopharyngeal carcinoma which is not amenable to curative treatment with surgery and/or radiation therapy.
* 2. Age ≥ 18 years and ≤ 75 years, both genders.
* 3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
* 4. Life expectancy of at least 3 months.
* 5. Have failed for first-line platinum-based chemotherapy.
* 6. Have failed for prior treatment with PD-1 antagonists +/- chemotherapy.
* 7. Patients must have at least 1 lesion that is measurable using RECIST v1.1 criteria.
* 8. Patients must have adequate organ function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment) as determined by: Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ 75×109/L; Hemoglobin ≥ 9 g/dL; serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN), (for subjects with liver metastases, TBIL ≤3×ULN ; ALT and AST≤5×ULN); Creatinine ≤1.5×ULN or creatinine clearance rate≥50 ml/min (Cockcroft-Gault formula); serum albumin ≥28 g/L; Thyroid-stimulating hormone (TSH) levels ≤1×ULN (however, patients with free Triiodothyronine [FT3] or free Thyroxine [FT4] levels ≤1× ULN may be enrolled); INR, APTT≤1.5 x ULN.
* 9. All women with fertility potential must undergo a urine or serum pregnancy test during screening and the results are negative.

  10. Written informed consent.

Exclusion Criteria:

* 1.Known history of hypersensitivity to any components of the Tislelizumab formulation, or other monoclonal antibody.
* 2.Prior therapy with any anti-interleukin-4 receptor α (IL-4Rα) monoclonal antibody, anti-IgE monoclonal antibody, or other monoclonal antibodies/biological agents.
* 3.There was a history of severe bleeding, and any bleeding events with a serious grade of 3 or more in CTCAE5.0 occurred within 4 weeks before screening.
* 4.Before treatment, MRI showed that the tumor may have invaded important blood vessels (such as enclosing the internal carotid artery / vein), nasopharyngeal necrosis, or researchers have determined that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during treatment.
* 5.Patients with abnormal blood coagulation and bleeding tendency (14 days before signing informed consent: INR is within the normal range without anticoagulant); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues. On the premise that the INR < 1.5, low-dose warfarin (1mg orally, once a day) or low-dose aspirin (daily dose not more than 100mg) is allowed for preventive purposes.
* 6.Arteriovenous thrombosis occurred within one year before screening, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis (except venous thrombosis caused by intravenous catheterization due to early chemotherapy) and pulmonary embolism.
* 7. Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as basal cell skin cancer or carcinoma in situ of the cervix.
* 8. Join another clinical study at the same time, received any research drug within 4 weeks before the first administration of the drug.
* 9. Patients with any active autoimmune disease or a documented history of autoimmune disease such as pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism;
* 10. Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids. Doses > 10 mg/day prednisone or equivalent are prohibited within 2 weeks before study drug administration.
* 11. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease.
* 12. Be known to have active tuberculosis.
* 13. Hepatitis B virus (HBV) >2000 IU/ml or DNA ≥ 1×10^4/ml; or hepatitis C virus (HCV) RNA ≥ 1×10^3/ml).
* 14. Has an active infection requiring systemic therapy.
* 15. Has known active central nervous system metastases.
* 16. Severe, uncontrolled angiocardiopathy (heart failure > class II NYHA, unstable angina, myocardial infarction within past 1 year, supraventricular or ventricular arrhythmia which need medical intervention, or QT interval male ≥ 450 ms, female ≥ 470 ms.).
* 17. Have been vaccinated with anti-tumor vaccines or have been vaccinated with live vaccines within 4 weeks before screening.
* 18. Pregnant or nursing.
* 19. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 2 years
  An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI)

SECONDARY OUTCOMES:
Disease control rate | 2 years
  A disease control rate is defined as either a confirmed CR or a PR or a SD, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI).
Duration of response | 2 years
  Defined from date of first confirmed CR or a PR to date of first documentation of progression or death due to any cause, as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI).
Progression-free survival rate | 2 years
  Defined from date of registration to date of first documentation of progression or death due to any cause.
Overall survival rate | 2 years
  Defined from date of registration to date of first documentation of death from any cause or censored at the date of the last follow-up.
Incidence rate of adverse events (AEs) | 2 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events (acute toxicity) as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Qin S, Chan SL, Gu S, Bai Y, Ren Z, Lin X, Chen Z, Jia W, Jin Y, Guo Y, Hu X, Meng Z, Liang J, Cheng Y, Xiong J, Ren H, Yang F, Li W, Chen Y, Zeng Y, Sultanbaev A, Pazgan-Simon M, Pisetska M, Melisi D, Ponomarenko D, Osypchuk Y, Sinielnikov I, Yang TS, Liang X, Chen C, Wang L, Cheng AL, Kaseb A, Vogel A; CARES-310 Study Group. Camrelizumab plus rivoceranib versus sorafenib as first-line therapy for unresectable hepatocellular carcinoma (CARES-310): a randomised, open-label, international phase 3 study. Lancet. 2023 Sep 30;402(10408):1133-1146. doi: 10.1016/S0140-6736(23)00961-3. Epub 2023 Jul 24. PMID 37499670
- [Result] Zhang Y, Yan B, Shen S, Song X, Jiang Y, Shi L, Zhao C, Yang Y, Jiang L, Li J, Ye J, Liu J, Wan L, Yang Y, Chen J, Liu F, Su L, Xu Y, Tan G, Yu S, Zhang Y, Wang L, Liu S, Yan H, Liu W, Chen B, Wang C, Zhang L. Efficacy and safety of CM310 in severe eosinophilic chronic rhinosinusitis with nasal polyps (CROWNS-1): a multicentre, randomised, double-blind, placebo-controlled phase 2 clinical trial. EClinicalMedicine. 2023 Jul 5;61:102076. doi: 10.1016/j.eclinm.2023.102076. eCollection 2023 Jul. PMID 37483544
- [Result] Ng WT, Lee MC, Chang AT, Chan OS, Chan LL, Cheung FY, Hung WM, Chan CC, Lee AW. The impact of dosimetric inadequacy on treatment outcome of nasopharyngeal carcinoma with IMRT. Oral Oncol. 2014 May;50(5):506-12. doi: 10.1016/j.oraloncology.2014.01.017. Epub 2014 Feb 13. PMID 24529762
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593